CLINICAL TRIAL: NCT05232123
Title: Cannabidiol Effects on Cardiovascular System and Exercise Responses
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: did not receive funding
Sponsor: Castleton University (Other)
Responsible Party: Principal Investigator, Andrea Corcoran, Assistant Professor of Exercise Science, Castleton University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: VBRN Project 2022_Corcoran
Record Dates: First submitted 2022-01-11; First posted 2022-02-09 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Each participant will receive a different dose in consecutive weeks (one of which is a placebo), thus serving as their own control.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants will ingest 3ml of non-CBD containing MCT (medium-chain triglycerides) oil.
  Interventions: Drug: Placebo
- Cannabidiol 25 mg (Experimental): Participants will ingest 3ml of MCT (medium-chain triglycerides) oil containing 25 mg of CBD.
  Interventions: Drug: Cannabidiol
- Cannabidiol 50 mg (Experimental): Participants will ingest 3ml of MCT (medium-chain triglycerides) oil containing 50 mg of CBD.
  Interventions: Drug: Cannabidiol
- Cannabidiol 200 mg (Experimental): Participants will ingest 3ml of MCT (medium-chain triglycerides) oil containing 200 mg of CBD.
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Placebo — Placebo oral product formulated in MCT (medium chain triglyceride) oil
  Arms: Placebo
Drug: Cannabidiol — Cannabidiol oral product formulated in MCT (medium chain triglyceride) oil
  Other Names: CBD
  Arms: Cannabidiol 200 mg; Cannabidiol 25 mg; Cannabidiol 50 mg

SUMMARY:
To identify the autonomic effects of recreationally-relevant doses of cannabidiol (CBD) in an older population, and to evaluate the effect of CBD on exercise performance and recovery.

DETAILED DESCRIPTION:
Heart rate variability (HRV) analysis is a common method used to evaluate the function of the autonomic nervous system. While heart rate is the number of heart beats per minute, HRV is the fluctuation of the time intervals between those beats (interbeat intervals). If the interbeat intervals are too similar, this is an indication of an unhealthy heart. A major influence on heart rate (and thus interbeat interval), is the autonomic nervous system which is divided into two branches: sympathetic and parasympathetic. HRV represents the balance between both systems, with higher HRV being associated with greater parasympathetic activity, and lower HRV with greater sympathetic activity. While there is no optimal level of HRV, a higher HRV is associated with reduced stress and good health, and a lower HRV is associated with chronic diseases and cardiovascular risk. The current study will evaluate the effect of recreationally-relevant doses of CBD (25-200mg) on resting HRV in older adults (aims 1&2). Investigators will also look at the effects of CBD on cardiovascular fitness by having participants complete a maximum graded exercise test under the influence of a placebo and again after ingesting a single dose of CBD (aims 3&4).

ELIGIBILITY:
Inclusion Criteria:

* male or female
* 18+ years (aims 3&4)
* 50+ years (aims 1&2)
* participants must agree to fast for 4 hours and abstain from food or beverages containing alcohol, caffeine, or CBD for 12 hours prior to each experimental session
* participants must agree to avoid exercise for 6 hours prior to each experimental session
* completion of Health History Screening Questionnaire with report indicating overall good health
* ability to comprehend and satisfactorily comply with protocol requirements
* written informed consent given prior to study participation
* low-risk for VO2max testing (aims 3&4)

Exclusion Criteria:

* women who are pregnant or lactating
* participants who have a history of adverse reactions to cannabidiol
* current medications that might influence the cardiovascular and/or autonomic systems
* any cardiac, pulmonary, renal, or metabolic disease
* walking difficulty (aims 3&4)
* waiting for a stress test for a medical reason (aims 3&4)
* medical contraindication to performing a treadmill stress test (aims 3&4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate variability (HRV) as assessed by time-domain analysis: standard deviation of RR intervals. | 4 weeks
  Time-domain measurements quantify the amount of variability of the heart's interbeat (RR) intervals and include the metric: standard deviation of RR intervals (SDNN). Higher values indicate greater HRV.
Change in heart rate variability (HRV) as assessed by time-domain analysis: root mean square of successive differences. | 4 weeks
  Time-domain measurements quantify the amount of variability of the heart's interbeat (RR) intervals and include the metric: root mean square of successive differences (RMSSD). Higher values indicate greater HRV.
Change in heart rate variability (HRV) as assessed by frequency-domain analysis: high-frequency (HF). | 4 weeks
  Frequency-domain measurements estimate the distribution of absolute or relative power into four heart rate oscillation frequency bands: ultra-low-frequency (ULF), very-low-frequency (VLF), low-frequency (LF) and high-frequency (HF). A high HF reflects parasympathetic dominance.
Change in heart rate variability (HRV) as assessed by frequency-domain analysis: low-frequency (LF). | 4 weeks
  Frequency-domain measurements estimate the distribution of absolute or relative power into four heart rate oscillation frequency bands: ultra-low-frequency (ULF), very-low-frequency (VLF), low-frequency (LF) and high-frequency (HF). LF reflects both sympathetic and parasympathetic activity.
Change in heart rate variability (HRV) as assessed by frequency-domain analysis: LF/HF ratio. | 4 weeks
  A low LF/HF ratio reflects parasympathetic dominance, whereas a high LF/HF ratio reflects sympathetic dominance.
Change in magnitude of autonomic stress test responses as assessed by changes in blood pressure. | Week 5
  Responses to autonomic stress test include a change in blood pressure if sympathetic outflow is activated. The magnitude of change will be compared before and after CBD ingestion.
Change in magnitude of autonomic stress test responses as assessed by changes in heart rate. | Week 5
  Responses to autonomic stress test include a change in heart rate if parasympathetic outflow is activated. The magnitude of change will be compared before and after CBD ingestion.
Maximal oxygen consumption (VO2max) | 8 days
  Maximum oxygen consumption will be calculated during treadmill test (using the Bruce Protocol)
Heart rate | through study completion, an average of 4 weeks
  Change in heart rate will be assessed throughout session

SECONDARY OUTCOMES:
Blood pressure | through study completion, an average of 4 weeks
  Change in blood pressure will be assessed throughout session
Borg's Category-Ratio Scale for Rating of Perceived Exertion | 8 days
  The Borg Scale is a self-reporting instrument assessing intensity of perceived exertion on a 0 to 10 scale, 0 being rest and 10 maximal effort.

OTHER OUTCOMES:
Change in oxygen saturation | 8 days
  percent O2 saturation measured by pulse oximeter throughout session
Blood lactate | 8 days
  Plasma lactate assess by finger stick
Change in exercise duration | 8 days
  Total exercise time on the treadmill while performing the Bruce Protocol.
Breathing frequency | 8 days
  Breathing frequency will be measured throughout session
Tidal volume | 8 days
  Tidal volume will be measured throughout session

CONTACTS AND LOCATIONS:
Locations (1):
- Castleton University, Jeffords Science Building, Castleton, Vermont, United States

IPD SHARING:
Plan to Share IPD: No